CLINICAL TRIAL: NCT01021306
Title: Conservative Treatment of Patients With Temporomandibular Disorders
Acronym: D1P2-TMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palmer College of Chiropractic (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); University of Iowa (Other); Schaeffer Chiropractic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DCRC1-P2; 5U19AT004663-02 (NIH)
Record Dates: First submitted 2009-11-24; First posted 2009-11-26 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-04

CONDITIONS: Temporomandibular Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Self Care; Dental Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Chiropractic w/Activator & Self Care (Active Comparator): This technique uses a hand held instrument to deliver a quick, shallow thrust in a well defined manner.
  Interventions: Device: Chiropractic w/Activator & Self Care
- Dental Care & Self Care (Active Comparator): Intraoral splints are removable orthopedic appliances fabricated of hard acrylic resin positioned between the remaining teeth of the patient. They are designed in theory to support the function of the TMJ and relieve associated pain. Stabilization splints are believed to function by stabilizing the intracapsular structure of the TMJ, reducing activity of masticatory muscles, distributing occlusal forces, and reducing bruxism (teeth grinding).
  Interventions: Device: Dental Care & Self Care
- Sham AMCT & Self Care (Sham Comparator): This protocol will attempt to follow all of the procedures of the actual AMCT protocol except no thrust will be delivered. Self-care only participants successfully completing the 6 month assessment will be given the option for RIST or AMCT for one month.
  Interventions: Other: Sham AMCT
- Self-care only group (Placebo Comparator): All patients will be offered the self-care checklist of homecare approaches at baseline. Self-care only participants successfully completing the 6 months assessment will be given the option for RIST or AMCT for one month.
  Interventions: Other: Self-Care Only Group

INTERVENTIONS:
Device: Chiropractic w/Activator & Self Care — This technique uses a hand held instrument to deliver a quick, shallow thrust in a well defined manner. The instrument has two handles that are squeezed together until it clicks, resulting in a shallow, very quick thrust to the segment that is to be adjusted. The AMCT protocol is a structured method of chiropractic treatment that utilized a number of simple biomechanical tests in order to determine where to adjust. These tests are mostly well defined movements of body parts such as extending the head or laterally moving the mandible relative to the rest of the skull. This protocol includes treatment of the full spine and appendages as well as the area immediately around the jaw.
  Arms: Chiropractic w/Activator & Self Care
Device: Dental Care & Self Care — Following the dental exam, patients will have maxillary and mandibular polyvinyl siloxane impressions made. Interocclusal records will be made with a fast setting silicone using a metal tray. A commercial laboratory will then wax and heat process a clear acrylic resin splint attempting to capture the mandibular cusp tips in the occlusal plan of the splint. The splint will be adjusted to provide uniform posterior centric occlusal stops followed by evaluation for canine guidance. The splint will then be polished and home care instruction provided. Patients will be instructed to wear the splint at night and two hours per day.
  Arms: Dental Care & Self Care
Other: Sham AMCT — This protocol will attempt to follow all of the procedures of the actual AMCT protocol except that when a thrust is given with the Activator instrument, the clinician will place the thumb of his left hand over the spot that would normally be adjusted. The tip of the instrument them will be placed very close to, but not touching the thumb. Consequently, the patient will feel the contact of the clinician's thumb on the spot that would be normally adjusted, and will hear the click of the instrument, but no thrust will be delivered to the patient.
  Arms: Sham AMCT & Self Care
Other: Self-Care Only Group — Self care consists of an initial set of standard patient self performed treatments which will include jaw relaxation exercises, reduction of parafunction, thermal packs, low dose NSAIDs, passive opening stretches and suggestions for stress reduction.
  Arms: Self-care only group

SUMMARY:
At any given time, 10 million Americans suffer from temporomandibular disorders (TMD), with a lifetime prevalence of 45% and costs for direct care exceeding $2 billion/year. Little evidence exists regarding the efficacy of specific conservative interventions used to treat TMD and currently there is no "gold standard" of care that is widely accepted by the dental or medical community. This study is a prospective, randomized 4 arm parallel observer-masked pilot study comparing: 1) Activator Methods Chiropractic Technique (AMCT), 2) a conservative dental approach with reversible interocclusal splint therapy, 3) a sham AMCT, and 4) a self-care only group, which includes a standard checklist of self-care jaw relaxation techniques, for a total of 80 patients with chronic myofascial TMD.

DETAILED DESCRIPTION:
All patients will be offered the self-care checklist of homecare approaches at baseline. Patients will be treated for two months with follow up at 3 and 6 months after enrollment. The primary outcome measure will be an 11 point Numerical Rating Scale for average TMD pain during the past week. Secondary outcomes will include the Oral Health Impact Profile (OHIP-14), believability of the sham AMCT compared to active AMCT, expectations of and satisfaction with care, medication use, bothersomeness of symptoms and health care utilization. Our project is a collaborative effort between the Palmer Center for Chiropractic Research (PCCR) and the University of Iowa (UI) through the College of Dentistry and the General Clinical Research Center (GCRC) Oral and Craniofacial Unit. The PCCR Clinic and Data Core will serve as the data coordinating center and will develop a web-based data collection system for this project. Patient eligibility will be assessed by dental examiners at the UI College of Dentistry using the Research Diagnostic Criteria for Temporomandibular Disorders to diagnose chronic, Axis I myofascial TMD. Dental care will be provided by a dentist at UI GCRC and chiropractic care will be provided by a private practitioner in close proximity to UI. The aims of this project are to assess the feasibility of conducting a full-scale randomized clinical trial to evaluate the effectiveness of AMCT for patients with chronic myofascial TMD; determine the most appropriate control group(s) for a full-scale randomized controlled trial; and to estimate the sample size needed for an adequately-powered trial and the recruitment period that would be required. In general, there is a lack of evidence for the efficacy of non-surgical treatment for patients with TMD, including chiropractic interventions. If the beneficial effects of the AMCT are supported in this pilot study, the logistical information gained will allow us to plan a full scale trial for patients suffering pain and disability due to TMD. It is anticipated that such a trial will allow clinicians to make more informed recommendations for treatment of patients with TMD. At the conclusion of this project, we will be well-positioned to prepare an R01 level grant application.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older
* TMD symptoms for at least 6 months
* Must have 7-8 teeth per dental arch that are in occlusion (can be restored teeth or dental implants with crowns or fixed dental bridgework)
* Typical TMD pain during the past week > = 3 on an 11 point Numerical Rating Scale
* RDC/TMD Axis I diagnosis of myofascial pain (Group Ia or Ib) with or without a concurrent diagnosis of arthralgia (Group IIIa) or disk displacement with reduction (Group IIa)
* Stable prescription medication plan: no changes in prescription medication for pain during the past month

Exclusion Criteria:

* Current or pending litigation for a personal injury case, worker's compensation, or disability
* Participants with unstable periodontitis and/or a dental condition with untreated disease (e.g., caries). Participants may elect to have her/his dental care provided to stabilize their dental condition prior to randomization.
* Subjects with Canine Class II malocclusion that would prohibit fabrication of RIST appliance
* Cases that need further diagnostic procedures to rule in or rule out the condition (i.e., MRI or CT scan)
* Systemic arthritis or other serious medical condition necessitating maximum daily dosing of COX-2 inhibitor or NSAIDs, (All NSAID use will be recorded in the daily diary as a part of the Self-Care data recording).
* Participants presenting with complete dentures
* Any treatment for TMD during the previous month, except for non-prescription medications or a stable prescription medication regimen for TMD.
* Inability to read or verbally comprehend English
* Unwillingness to be enrolled in any of the four intervention groups.
* Unwillingness to postpone other forms of treatment for TMD during the two month active care phase (except for non-prescription medications or continuation of a stable prescription medication regimen).
* Unwillingness to postpone any chiropractic care during the two month active care phase.
* Intention to move from the area during the next seven months
* Ever had active chiropractor care for TMD pain
* Drug or alcohol abuse
* Pregnant or planning to be pregnant during next seven months
* MVA or other trauma in the last six months
* Facial pain/TMD not worst pain
* General poor health
* Extensive dental work in past 6 months including orthodontics
* Serious co-morbid conditions, including: Lupus Erythematosus, Sjogren's Syndrome, Multiple Sclerosis, Symptomatic Trigeminal Neuralgia (tic/tic douloureux) or any other neuralgia of the face, Thyroid problem not controlled by medication, Uncontrolled diabetes, Rheumatoid arthritis, Fibromyalgia, Polymyalgia Rheumatic, Giant Cell Arteritis, Psoriatic Arthritis, Reiters Syndrome, Bechets Syndrome, Crohn's Disease, Ulcerative Colitis, Parkinson's Disease, Tardive Dyskinesia, Active seizure disorder, Stroke with head and neck symptoms, Addison's Disease, Cushing's Disease
* Have had or ever had any type of head or neck surgery within the last 6 months
* Have had or ever had radiation treatment to the head and/or neck
* Have had or ever had surgery of your jaw joints, not including arthroscopic surgery
* Have had or ever had Herpes Zoster or shingles in the face

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James W DeVocht, DC, PhD, Principal Investigator — Palmer College of Chiropractic
Locations (3):
- United States (3):
  - Schaeffer Chiropractic, Coralville, Iowa
  - Palmer College of Chirpractic, Davenport, Iowa
  - University of Iowa College of Dentistry, Iowa City, Iowa

IPD SHARING:
Plan to Share IPD: Yes
Once the resulting manuscripts have been published, data sets will be provided for public access. Potential investigators can contact one of the Co-PIs to present their hypothesis, study design, instruments and/or data on which to focus, and resources required. Depending upon the needs and desires of the requesting party, the data that are shared may include analytic tables or de-identified or limited data sets that are transmitted to the requesting parties for additional analyses.

REFERENCES:
- [Background] Salsbury SA, DeVocht JW, Hondras MA, Seidman MB, Stanford CM, Goertz CM. Chiropractor interaction and treatment equivalence in a pilot randomized controlled trial: an observational analysis of clinical encounter video-recordings. Chiropr Man Therap. 2014 Dec 3;22(1):42. doi: 10.1186/s12998-014-0042-7. eCollection 2014. PMID 25478142
- [Background] Dodes JE. More about chiropractics. J Am Dent Assoc. 2014 Feb;145(2):127. doi: 10.1016/s0002-8177(14)60212-9. No abstract available. PMID 24487602
- [Background] Digregorio CJ. Questioning chiropractics. J Am Dent Assoc. 2014 Feb;145(2):127. doi: 10.1016/s0002-8177(14)60211-7. No abstract available. PMID 24487601
- [Background] Glick M, Pihlstrom BL. Response from the JADA Editor and the Associate Editor, Research. J Am Dent Assoc. 2014 Feb;145(2):127-8. doi: 10.1016/s0002-8177(14)60213-0. No abstract available. PMID 24487603
- [Result] DeVocht JW, Goertz CM, Hondras MA, Long CR, Schaeffer W, Thomann L, Spector M, Stanford CM. A pilot study of a chiropractic intervention for management of chronic myofascial temporomandibular disorder. J Am Dent Assoc. 2013;144(10):1154-63. doi: 10.14219/jada.archive.2013.0034. PMID 24080932

RESULTS

PARTICIPANT FLOW:
Groups:
- Dental Care & Self Care: Intraoral splints are removable orthopedic appliances made of acrylic resin positioned between remaining teeth and designed in theory to support function of the TMJ and relieve pain. Stabilization splints are believed to function by stabilizing intracapsular structure of TMJ, reducing activity of masticatory muscles, distributing occlusal forces, and reducing bruxism (teeth grinding).
  Dental Care & Self Care: Following dental exam, patients will have maxillary and mandibular polyvinyl siloxane impressions. Interocclusal records will be made with a fast setting silicone using a metal tray. Commercial laboratory will wax and heat process acrylic resin splint to capture mandibular cusp tips in the occlusal plan of splint. Splint will be adjusted to provide uniform posterior centric occlusal stops followed by evaluation for canine guidance. Splint will be polished and home care instruction provided. Patients will be i
Period: 2 Month (Primary Outcome)
Arm/Group | Chiropractic w/Activator & Self Care | Dental Care & Self Care | Sham AMCT & Self Care | Self-care Only Group
Started | 20 | 20 | 19 | 21
Completed | 14 | 14 | 14 | 17
Not Completed | 6 | 6 | 5 | 4
Period: 6 Month (Follow-up)
Arm/Group | Chiropractic w/Activator & Self Care | Dental Care & Self Care | Sham AMCT & Self Care | Self-care Only Group
Started | 14 | 14 | 14 | 17
Completed | 11 | 13 | 14 | 14
Not Completed | 3 | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chiropractic w/Activator & Self Care | Dental Care & Self Care | Sham AMCT & Self Care | Self-care Only Group | Total
Number analyzed (Participants) | 20 | 20 | 19 | 21 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (7.9) | 36.9 (13.5) | 33.1 (11.4) | 38.0 (12.7) | 35.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 15 | 16 | 64
  Male | 4 | 3 | 4 | 5 | 16
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 19 | 21 | 80

OUTCOME MEASURES:

1. Primary Outcome: Patient-Rated TMD Pain, an 11 Point Numerical Rating Scale (NRS)
Description: The Numerical Rating Scale ranges from 0 (no pain) to 10 (pain as bad as it can be).
Time Frame: 2 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Chiropractic w/Activator & Self Care | Dental Care & Self Care | Sham AMCT & Self Care | Self-care Only Group
Number analyzed (Participants) | 20 | 20 | 19 | 21
units on a scale | 0.9 [-0.1 to 1.8] | 1.4 [0.3 to 2.5] | 1.6 [0.6 to 2.6] | 0.7 [-0.1 to 1.5]

2. Secondary Outcome: Oral Health Impact Profile (OHIP-14)
Description: The OHIP-14 contains 2 questions about each of 7 dimensions (14 items), indicating how often the participant had experienced each difficulty in the previous month; possible responses range from 0 (never) to 4 (very often). The OHIP score was obtained by summing the 14 ratings.
Time Frame: 2 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Chiropractic w/Activator & Self Care | Dental Care & Self Care | Sham AMCT & Self Care | Self-care Only Group
Number analyzed (Participants) | 20 | 20 | 19 | 21
units on a scale | 1.3 [-2.3 to 5.0] | 3.6 [0.1 to 7.2] | 2.0 [-1.8 to 5.8] | 2.8 [-0.4 to 6.1]

3. Secondary Outcome: Bothersomeness of Symptoms
Description: Possible ratings range from 1 (not at all bothersome) to 5 (extremely bothersome)
Time Frame: 2 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Chiropractic w/Activator & Self Care | Dental Care & Self Care | Sham AMCT & Self Care | Self-care Only Group
Number analyzed (Participants) | 20 | 20 | 19 | 21
units on a scale | 2.3 [0.5 to 4.1] | 2.4 [0.6 to 4.2] | 2.3 [0.7 to 4.0] | 1.8 [0.3 to 3.3]

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Chiropractic w/Activator & Self Care | Dental Care & Self Care | Sham AMCT & Self Care | Self-care Only Group
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/19 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No